CLINICAL TRIAL: NCT01909440
Title: Exercise and Protein Supplementation for Prostate Cancer Survivors Receiving Androgen Deprivation Therapy
Brief Title: Resistance Training and Protein Supplementation for Prostate Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4P-13-2; NCI-2013-01360 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-13-00315; P30CA014089 (NIH)
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (RT + PS) (Experimental): Patients undergo total body high-intensity RT thrice weekly and perform static stretching exercises after each session. Exercises progress from low intensity and high volume to higher intensity and lower volume over the course of the 12-week program. Patients also receive whey protein supplementation orally twice a day for 12 weeks.
  Interventions: Behavioral: exercise intervention; Dietary Supplement: nutritional supplementation; Procedure: quality-of-life assessment; Other: questionnaire administration; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (total body RT) (Experimental): Patients undergo total body RT and stretching as in Arm I.
  Interventions: Behavioral: exercise intervention; Procedure: quality-of-life assessment; Other: questionnaire administration; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm III (protein supplementation) (Experimental): Patients receive whey protein supplementation as in Arm I. Patients also undergo a home flexibility program 3 times per week, consisting of the same static stretching exercises performed after RT. After 12 weeks, patients may undergo the RT program as in Arm I.
  Interventions: Dietary Supplement: nutritional supplementation; Procedure: quality-of-life assessment; Other: questionnaire administration; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm IV (attention control) (Active Comparator): Patients undergo the home flexibility program as in Arm III. After 12 weeks, patients may undergo total body RT as in Arm I.
  Interventions: Procedure: quality-of-life assessment; Other: questionnaire administration; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Behavioral: exercise intervention — Receive whole body RT
  Arms: Arm I (RT + PS); Arm II (total body RT)
Dietary Supplement: nutritional supplementation — Given whey protein supplementation PO
  Arms: Arm I (RT + PS); Arm III (protein supplementation)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot clinical trial studies resistance training and protein supplementation in increasing lean body mass in patients with prostate cancer receiving androgen deprivation therapy. Resistance training and protein supplementation may help improve quality of life in patients with prostate cancer receiving androgen deprivation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the effects of progressive, structured resistance training (RT) program , with and without protein supplementation (PS), on lean body mass (LBM) in prostate cancer survivors (PCS) on androgen deprivation therapy (ADT). Increases in LBM may influence additional outcomes such as physical function, quality of life (QOL) and molecular pathways that regulate skeletal muscle.

SECONDARY OBJECTIVES:

I. To examine the effects of a structured RT program, with and without PS, on muscle strength, physical function, and QOL in PCS on ADT .

TERTIARY OBJECTIVES:

I. To examine the effects of a progressive, structured RT program, with and without PS, on anabolic and catabolic molecular regulators of skeletal muscle in PCS on ADT.

II. To examine the effects of a progressive, structured RT program, with and without PS, on bone turnover markers and bone mineral density in PCS on ADT.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients undergo total body high-intensity RT thrice weekly, and perform static stretching exercises after each session. Exercises progress from low intensity and high volume to higher intensity and lower volume over the course of the 12-week program. Patients also receive whey protein supplementation orally twice a day for 12 weeks.

ARM II: Patients undergo total body RT and stretching as in Arm I.

ARM III: Patients receive whey protein supplementation as in Arm I. Patients also undergo a home flexibility program 3 times per week, consisting of the same static stretching exercises performed after RT. After 12 weeks, may undergo the RT program as in Arm 1.

ARM IV: Patients undergo the home flexibility program as in Arm III. After 12 weeks, patient may undergo total body RT as in Arm 1.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer

  * Treatment with androgen deprivation therapy (ADT) (gonadotropin-releasing hormone [GnRH] agonist/antagonist with or without anti-androgen) for prostate cancer
  * Receiving ADT for a minimum of 12 weeks before enrollment into the study
  * Planned ADT for the duration of the 12-week study period
* Asymptomatic, or minimally symptomatic from prostate cancer or prostate cancer related therapies

  * No opioid-requiring cancer related pain
  * Any therapy related genitourinary or gastrointestinal symptoms should be considered as mild (Common Terminology Criteria for Adverse Events [CTCAE] grade 1 or 2) and not interfering with activities of daily living
* Permission from treating/study physician to participate in RT

Exclusion Criteria:

* No concurrent use of chemotherapy or radiotherapy (radiotherapy should be completed at least 4 weeks from study entry)
* History of allergic reactions to whey protein
* Milk protein intolerance/allergies (lactose intolerance is acceptable)
* Subjects currently using N-acetylcysteine, alpha-lipoic acid supplements, or dry whey protein supplements
* Recovered from major surgery within the last 6 months
* Acute coronary (e.g. myocardial infarction) or vascular event within the last year as well as uncontrolled coronary heart disease (e.g. progressive angina)
* Stroke within the past 2 years
* Neurologic and/or orthopedic limitations that preclude the participation in the training program (e.g. bone metastases that may pose a high risk of pathologic fracture)
* Subjects currently participating in a RT program

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Completion of the resistance training program with at least 80% of the sessions attended | 12 weeks
Compliance with protein supplementation | 12 weeks
Change in lean body mass | Baseline up to 12 weeks
  Intent-to-treat models will be computed using repeated measures analysis of variance (ANOVA).
Change in strength | Baseline up to 12 weeks
  Intent-to-treat models will be computed using repeated measures ANOVA.
Change in quality of life | Baseline up to 12 weeks
  Intent-to-treat models will be computed using repeated measures ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: E. Todd Schroeder, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Dawson JK, Dorff TB, Tuzon C, Rice JC, Schroeder ET, Lane CJ, Gross ME, Dieli-Conwright CM. Effect of Periodized Resistance Training on Skeletal Muscle During Androgen Deprivation Therapy for Prostate Cancer: A Pilot Randomized Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211035442. doi: 10.1177/15347354211035442. PMID 34301165
- [Derived] Dawson JK, Dorff TB, Todd Schroeder E, Lane CJ, Gross ME, Dieli-Conwright CM. Impact of resistance training on body composition and metabolic syndrome variables during androgen deprivation therapy for prostate cancer: a pilot randomized controlled trial. BMC Cancer. 2018 Apr 3;18(1):368. doi: 10.1186/s12885-018-4306-9. PMID 29614993
- [Derived] Kiwata JL, Dorff TB, Todd Schroeder E, Salem GJ, Lane CJ, Rice JC, Gross ME, Dieli-Conwright CM. A pilot randomised controlled trial of a periodised resistance training and protein supplementation intervention in prostate cancer survivors on androgen deprivation therapy. BMJ Open. 2017 Jul 10;7(7):e016910. doi: 10.1136/bmjopen-2017-016910. PMID 28698349